CLINICAL TRIAL: NCT01325194
Title: Dose Densified Chemoimmunotherapy With Early CNS Prophylaxis in Patients Less Than 65 Years With High Risk (aaIPI≥ 2) Diffuse Large B-Cell Lymphoma
Brief Title: CHemoImmunotherapy With Early Central Nervous System (CNS) Prophylaxis
Acronym: CHIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Lymphoma Group (Network)
Collaborators: Mundipharma Pte Ltd. (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG-LBC-05
Record Dates: First submitted 2011-03-14; First posted 2011-03-29 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Primary Disease
Keywords: DLBCL; FL grade 3B; high risk; CNS prophylaxis; chemoimmunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CNS prophylaxis (Experimental)
  Interventions: Drug: liposomal cytarabine

INTERVENTIONS:
Drug: liposomal cytarabine — 50 mg intrathecally three times
  Other Names: Depocyte

SUMMARY:
The purpose is to test whether early central nervous system (CNS) prophylaxis given at the beginning of therapy for young high risk diffuse large B-cell lymphoma (DLBCL) patients is feasible and could reduce the risk of CNS relapses. Early CNS prophylaxis with two courses high dose methotrexate (HD-MTX) in combination with rituximab-cyclophosphamide-doxorubicin-vincristine-prednison (R-CHOP) is followed by four courses of R-CHOP14 and etoposide (E) and one course of HD-Ara-C. In addition the patients will receive three courses of liposomal cytarabine intrathecally. The results will be compared to a recent Nordic CRY-04 study. Shifting of CNS prophylaxis to the beginning of the therapy offers a potential to overcome the subclinical disease and thus reduce the risk of early clinical CNS recurrence. As flow cytometry (FCM) can improve the sensitivity for detecting occult leptomeningeal disease over cytology , FCM from cerebrospinal fluid will be incorporated into the staging procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 - < 65 years. Histologically confirmed CD20+ diffuse large B-cell lymphoma (DLBCL) based on WHO 2008 Lymphoma Classification
* Follicular lymphomas (FLs) grade 3b is allowed

Patients in at least stage II with age adjusted international prognostic score (IPI score) of 2 or 3:

* Stage III /IV and elevated LDH
* Stage III/IV and WHO performance status 2 - 3
* Stage II and elevated LDH and WHO performance status 2 - 3 And/or patients with
* More than one extranodal site
* Testicular lymphoma, stage IIE and higher
* Paranasal sinus and orbital lymphoma with destruction of bone
* Large cell infiltration of the bone marrow

Exclusion Criteria:

* Severe cardiac disease: cardiac function grade 3-4
* Impaired liver, renal or other organ function not caused by lymphoma, which will interfere with the treatment schedule
* Pregnancy/lactation
* Men and women of reproductive potential not agreeing to use an acceptable method of birth control during treatment and for six months after completion of treatment
* Patients with other severe medical problems and with an expected short survival for non-lymphoma reasons
* Known HIV positivity
* Uncontrolled infectious disease, including meningeal infection
* Active cancer except basal cell carcinoma and cervical carcinoma in situ during the last five years
* Earlier treatment containing anthracyclins
* Psychiatric or mental disorder which make the patient unable to give an informed consent and/or adhere to the protocol
* CNS disease as diagnosed by MRI or cerebrospinal fluid (CSF) cytology. Positive CSF flow cytometry below diagnostic threshold level by cytology is allowed
* Pleural or peritoneal fluid that cannot be drained safely
* Hypersensitivity to the active substance or any of the other ingredients
* Patients participating in other clinical studies, unless followed for survival

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure | 3 and 5 years

SECONDARY OUTCOMES:
Maximal hematological, gastrointestinal, neuronal and other toxicities | Treatment period (5 years)
Clinical response rate | Treatment period (5 years)
Incidence of central nervous system(CNS) relapse in cerebrospinal fluid (CSF )cytology neg/flow cytometry positive cases | 3 and 5 years
Incidence of CNS relapse in a subgroup of patients with more than one extranodal site and elevated lactate dehydrogenase (LDH) | 3 and 5 years
Progression free survival | 3 and 5 years
Overall survival | 3 and 5 years
Molecular predictors | 3 years
CNS relapse rate | 1,5 years

CONTACTS AND LOCATIONS:
Locations (4):
- Department of Hematology, Århus University Hospital, Aarhus, Denmark
- Department of Oncology, Helsinki University Central Hospital, Helsinki, Finland
- Department of Oncology, Oslo University Hospital, Oslo, Norway
- Department of Oncology, Lund University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Arffman M, Meriranta L, Autio M, Holte H, Jorgensen J, Brown P, Jyrkkio S, Jerkeman M, Drott K, Fluge O, Bjorkholm M, Karjalainen-Lindsberg ML, Beiske K, Pedersen MO, Leivonen SK, Leppa S. Inflammatory and subtype-dependent serum protein signatures predict survival beyond the ctDNA in aggressive B cell lymphomas. Med. 2024 Jun 14;5(6):583-602.e5. doi: 10.1016/j.medj.2024.03.007. Epub 2024 Apr 4. PMID 38579729
- [Derived] Vajavaara H, Leivonen SK, Jorgensen J, Holte H, Leppa S. Low lymphocyte-to-monocyte ratio predicts poor outcome in high-risk aggressive large B-cell lymphoma. EJHaem. 2022 Jun 23;3(3):681-687. doi: 10.1002/jha2.409. eCollection 2022 Aug. PMID 36051040
- [Derived] Leppa S, Jorgensen J, Tierens A, Meriranta L, Ostlie I, de Nully Brown P, Fagerli UM, Larsen TS, Mannisto S, Munksgaard L, Maisenholder M, Vasala K, Meyer P, Jerkeman M, Bjorkholm M, Fluge O, Jyrkkio S, Liestol K, Ralfkiaer E, Spetalen S, Beiske K, Karjalainen-Lindsberg ML, Holte H. Patients with high-risk DLBCL benefit from dose-dense immunochemotherapy combined with early systemic CNS prophylaxis. Blood Adv. 2020 May 12;4(9):1906-1915. doi: 10.1182/bloodadvances.2020001518. PMID 32380536
- [Derived] Autio M, Leivonen SK, Bruck O, Mustjoki S, Meszaros Jorgensen J, Karjalainen-Lindsberg ML, Beiske K, Holte H, Pellinen T, Leppa S. Immune cell constitution in the tumor microenvironment predicts the outcome in diffuse large B-cell lymphoma. Haematologica. 2021 Mar 1;106(3):718-729. doi: 10.3324/haematol.2019.243626. PMID 32079690
- See also: Related Info — http://www.nordic-lymphoma.org/